CLINICAL TRIAL: NCT03065478
Title: An Observational STudy to Evaluate the EFfectiveness of OnLife® in Improving Chemotherapy-induced peripherAl NeurOpathy in Patients With Colon or Breast Cancer After End of Adjuvant Therapy
Brief Title: Observational STudy to Evaluate the EFfectiveness of OnLife® in Improving CIPN in Patients With Colon or Breast Cancer After End of Adj. Therapy
Acronym: STEFANO
Status: Completed | Type: Observational
Sponsor: Swiss Medical Food AG (Industry)
Collaborators: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-080353
Record Dates: First submitted 2017-02-16; First posted 2017-02-28 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: CIPN in Adjuvant Colon Cancer Patients; CIPN in Adjuvant Breast Cancer Patients
Keywords: Peripheral Neuropathy; Chemotherapy induced; CIPN
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colon carcinoma: Dietary supplementation with "OnLife" to improve signs and symptoms of CIPN in adult colon cancer patients who experienced a CIPN after adjuvant oxaliplatin-containing chemotherapy.
  Interventions: Dietary Supplement: OnLife
- Mamma carcinoma: Dietary supplementation with "OnLife" to improve signs and symptoms of CIPN in adult breast cancer patients who experienced a CIPN after adjuvant paclitaxel regimen.
  Interventions: Dietary Supplement: OnLife

INTERVENTIONS:
Dietary Supplement: OnLife — Daily dosing of dietary supplement OnLife

SUMMARY:
The objective of this observational study is to evaluate the effectiveness of the dietary supplementation "OnLife" in improving signs and symptoms of chemotherapy-induced peripheral neuropathy (CIPN) in adult patients who have finished adjuvant oxaliplatin-containing regimen (colon cancer) or adjuvant paclitaxel regimen (breast cancer). Furthermore, patient-reported outcomes (PROs) and concomitant medication used for the treatment of neuropathic pain will be assessed.

DETAILED DESCRIPTION:
CIPN is a common side effect of many chemotherapeutic agents and often results in dose limitation, switch to less efficacious agents or even therapy discontinuation. CIPN mainly affects sensory nerves, while motor or autonomic nerve injury is rare. Therefore, most patients with CIPN experience numbness, tingling, hyperesthesia, loss of vibratory perception, and burning pain. Due to the vulnerability of the long nerves, CIPN typically appears in a 'stocking and glove' distribution.

Chemotherapeutic agents that cause CIPN include platinum compounds (e.g., cisplatin, oxaliplatin), antitubulins (vinca alkaloids (e.g., vincristine) and taxanes (e.g., docetaxel, paclitaxel)), proteasome inhibitors (e.g., bortezomib) and immunomodulatory drugs (e.g., lenalidomide).

Platinum compounds are known to accumulate in the dorsal root ganglion (DRG) leading to cell death in sensory neurons. DRG death may account for chronic sensory neuropathy, which manifests primarily as sensory paresthesias, dysesthesias and sensory ataxia most often located in the extremities and persists between cycles. In addition, Oxaliplatin directly regulates the gating of axonal voltage-gated sodium channels, inducing an acute neurotoxicity which is characterized by peripheral nerve hyperexcitability. Symptoms, like sensitivities to touching cold items, discomfort swallowing cold liquids, throat discomfort, and muscle cramps, occur during or shortly after the infusion.

Taxanes are known to cause disruption of microtubule function and therefore microtubule-based axonal transport. In addition, they interfere with macrophage activation in both the DRG and peripheral nerve, as well as microglial activation within the spinal cord. These effects result in a distal axonopathy also referred to as the dying-back phenomenon.

The effectiveness of OnLife® in improving CIPN is based on a patented fatty acid group (FAG) that comprises palmitoylethanolamide (PEA), alpha-linolenic acid, eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA), linoleic acid, oleic acid, palmitic acid, stearic acid, arachidic acid and myristic acid.

PEA, one main component of OnLife®, is an endogenous fatty acid amide belonging to the class of endocannabinoids and has been shown to have anti-inflammatory, antinociceptive, neuroprotective and anticonvulsant properties. It is synthesized in response to several inflammatory and painful disorders (e.g., intestinal inflammation and neuropathic pain) in order to counteract these pathological states. Clinical research revealed that treatment with exogenous PEA is effective and safe in various neuropathological conditions, including chronic idiopathic axonal neuropathy, diabetic neuropathy, nerve compression syndromes, as well as chemotherapy-induced neuropathic pain.

PEA exerts its analgesic and anti-inflammatory functions in the peripheral nervous system through its action on sensory neurons and on non-neuronal cells involved in inflammation, such as mast cells and macrophages. It indirectly activates cannabinoid receptor signaling by inhibiting the hydrolysis of endocannabinoids. This suppresses nociceptive behaviors and counteracts macrophage and mast cell activation, thereby reducing pain and other inflammatory symptoms. Another biological target of PEA is the nuclear peroxisome proliferator-activated receptor (PPAR)-alpha, expressed in various cells implicated in peripheral nociception, including dorsal DRG neurons and macrophages. Binding of PEA to PPAR-alpha ultimately results in reduced transcription of pro-inflammatory genes (e.g., TNF-alpha, IL-6, COX-2, iNOS) as well as repressed activity of pro-inflammatory transcription factors. In addition, there is some evidence that binding of PEA to PPAR-alpha may modulate excitability of primary sensory neurons by direct and indirect mechanisms.

The other fatty acids included in OnLife® have also been shown to have anti-inflammatory properties.

Currently, a study evaluating the efficacy and safety of OnLife® in patients with CIPN is carried out at the St. Savvas Anticancer Hospital, Athens by Dr. J. Skarlatos. First results suggest that OnLife® is reducing pain, numbness and tingle and improving heat/cold sensitivity as assessed by the physician. PRO, using the DN4 (Douleur Neuropathique 4) questionnaire, revealed a reduction of the score for diagnosing neuropathic pain during OnLife® application. Moreover, no patient showed a product-related side effect (date on file, unpublished).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with colon or breast cancer that have finished adjuvant oxaliplatin-containing or paclitaxel chemotherapy, respectively
* End of adjuvant chemotherapy does not date back more than 4 months
* Presence of CIPN grade 1-3 (according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.03)
* Decision for treatment with OnLife® (Baseline assessment has to be done before first intake of OnLife®)
* Written informed consent
* Able to understand and willing to complete study and patient-reported assessment instruments

Exclusion Criteria:

* Presence of sensory and/or motor disturbances due to other neurological diseases
* Alcohol abuse
* Pregnancy or breast-feeding
* Severe difficulty swallowing
* Intolerance to one of the ingredients of OnLife®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2 x 75 adult patients will be included. Cohort A: Adult patients with colon cancer who experience CIPN after end of adjuvant oxaliplatin-containing chemotherapy; Cohort B: Adult patients with breast cancer who experience CIPN after end of adjuvant paclitaxel chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the CIPN | 16 month
  Incidence of grade 0/1/2/3/4 peripheral sensory and/ or motor neuropathy according to CTCAE v4.03 after end of adjuvant oxaliplatin-containing regimen (colon cancer) or adjuvant paclitaxel regimen (breast cancer)

SECONDARY OUTCOMES:
Patient reported outcome: EORTC QLQ-C30 | 16 month
  Questionnaire EORTC QLQ-C30 is used to determine patients' health-related quality of life.
Patient reported outcome: EORTC QLQ-CIPN20 | 16 month
  Questionnaire EORTC QLQ-CIPN20 is used to elicit patients' experience of symptoms and functional limitations related to CIPN.
Concomitant medication used for the treatment of neuropathic pain | 16 month
  Drug treatment of neuropathic pain is observed over the time of the OnLife® application and the month after the end of OnLife® application

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Zaiss, Dr., Principal Investigator — Praxis für interdisziplinäre Onkologie & Hämatologie
Locations (1):
- Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No